CLINICAL TRIAL: NCT01906983
Title: Evaluation of Portal Venous System Thrombosis After Blunt Splenic Trauma Utilizing Doppler Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0159-13-RMBCTIL
Record Dates: First submitted 2013-06-23; First posted 2013-07-24 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Thrombosis of Portal Venous System.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Doppler ultrasound.: Doppler ultrasound will be performed to All patients 18 and up, admitted to Rambam Medical Center with diagnosis of blunt splenic trauma and agree to participate the study.
  Interventions: Other: Doppler Ultrasound

INTERVENTIONS:
Other: Doppler Ultrasound — Doppler ultrasound will be performed to patients with blunt splenic trauma, prior to discharge and again, at 3-6 months in patients with thrombosis indication.

SUMMARY:
The true incidence of thrombosis in the portal venous system after blunt splenic trauma is unknown and has not been elucidated in the medical literature. The investigators hypothesize that this entity is more common than previously suspected. Consequences of missing this diagnosis can be clinically significant, i.e. mesenteric ischemia in the acute phase and portal venous hypertension in the chronic phase. Early diagnosis would facilitate treatment with anticoagulation and avoidance of these complications. In a prospective fashion, doppler ultrasound will be performed prior to discharge and at 3 months in all patients 18 and up who have sustained blunt splenic trauma. Clinical follow-up will be extended to 6 months in patients initially diagnosed with thrombosis in the portal venous system on their 3 month ultrasound. The investigators will attempt to identify risk factors in this trauma population that would facilitate an early screening protocol.

ELIGIBILITY:
Inclusion Criteria:

* All trauma patients 18 and up admitted to Rambam Medical Center with diagnosis of blunt splenic trauma.

Exclusion Criteria:

* Trauma patients younger than 18.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All trauma patients 18 and up admitted to Rambam Medical Center with diagnosis of blunt splenic trauma.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Utilizing doppler ultrasound to assess the presence of partial or complete thrombosis in the portal venous system (splenic vein, superior mesenteric vein, inferior mesenteric vein and/or portal vein) after blunt splenic trauma. | Prior to discharge.

SECONDARY OUTCOMES:
Utilizing follow-up doppler ultrasound to assess change in the presence of partial or complete thrombosis in the portal venous system (splenic vein, superior mesenteric vein, inferior mesenteric vein and/or portal vein) after blunt splenic trauma. | 3 months following injury.

CONTACTS AND LOCATIONS:
Overall Officials: Hany Bahouth, M.D, Principal Investigator — Rambam Health Care Campus Haifa Israel
Locations (1):
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Background] Rajkomar V, Kyerematen E, Mysore P, Penston J. Thrombosis of the portal venous system following blunt abdominal trauma. BMJ Case Rep. 2010 Aug 24;2010:bcr1120092429. doi: 10.1136/bcr.11.2009.2429. PMID 22767370
- [Background] Fried M, Van Ganse W, Van Avermaet S. Mesenteric vein thrombosis triggered by blunt abdominal trauma in a patient with the primary antiphospholipid syndrome. Eur J Gastroenterol Hepatol. 2002 Jun;14(6):697-700. doi: 10.1097/00042737-200206000-00017. PMID 12072606
- [Background] Gonzalez F, Condat B, Deltenre P, Mathurin P, Paris JC, Dharancy S. Extensive portal vein thrombosis related to abdominal trauma. Gastroenterol Clin Biol. 2006 Feb;30(2):314-6. doi: 10.1016/s0399-8320(06)73173-6. PMID 16565670
- [Background] Gopal SV, Smith I, Malka V. Acute portal venous thrombosis after blunt abdominal trauma. Am J Emerg Med. 2009 Mar;27(3):372.e1-372.e3. doi: 10.1016/j.ajem.2008.07.021. No abstract available. PMID 19328396
- [Background] Beaufort P, Perney P, Coste F, Masbou J, Le Bricquir Y, Blanc F. [Post-traumatic thrombosis of the portal vein]. Presse Med. 1996 Feb 17;25(6):247-8. French. PMID 8729327
- [Background] Duvoux C, Radier C, Gouault-Heilmann M, Texier JP, Le Cudonnec B, Dhumeaux D. [A rare cause of portal vein thrombosis: closed abdominal trauma]. Gastroenterol Clin Biol. 1994;18(2):165-7. French. PMID 8013799
- [Background] Tran T, Demyttenaere SV, Polyhronopoulos G, Seguin C, Artho GP, Kaneva P, Fried GM, Feldman LS. Recommended timing for surveillance ultrasonography to diagnose portal splenic vein thrombosis after laparoscopic splenectomy. Surg Endosc. 2010 Jul;24(7):1670-8. doi: 10.1007/s00464-009-0828-1. Epub 2009 Dec 29. PMID 20039066